CLINICAL TRIAL: NCT05385653
Title: Pre-therapeutic Validation of the VR-based Exposure Scenario for CBT "ReVBEB" for the Induction of Food Craving in Patients With Bulimia and Binge Eating Disorder
Brief Title: Pre-therapeutic Validation of the Virtual Reality-based Exposure Scenario for CBT "ReVBED" for the Induction of Food Craving in Patients With Bulimia and Binge Eating Disorder (BED)
Acronym: RevBED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21CH086; ANSM (Other: 2021-A02307-34)
Record Dates: First submitted 2022-05-02; First posted 2022-05-23 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2023-11

CONDITIONS: Bulimia Nervosa; Binge-Eating Disorder
Keywords: food craving; virtual reality; eating disorders; bulimia nervosa; binge eating disorder
MeSH Terms: conditions — Bulimia Nervosa; Binge-Eating Disorder; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Cross-sectional, single-center comparative study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with bulimia or binge eating disorder (Experimental): patients with bulimia or binge eating disorder
  Interventions: Behavioral: experimentation of the virtual reality "RevBED"
- control (Other): paired healthy controls
  Interventions: Behavioral: experimentation of the virtual reality "RevBED"

INTERVENTIONS:
Behavioral: experimentation of the virtual reality "RevBED" — ReVBED is a VR-based exposure scenario for CBT for the induction of food craving in patients with bulimia nervosa and binge eating disorder.
  The use of ReVBED requires no VR experience and only generic and commonly used virtual reality tools (a computer with VR software, a wireless virtual reality headset, two controllers and headphones), all with a CE mark, allowing its users to move in and interact with a specially designed virtual environment.
  This exhibit scenario takes place in a VR environment built to represent a standard apartment consisting of four exhibit rooms (a bedroom, a teenager's bedroom, a living room and a kitchen) in which the ReVBED user moves sequentially through the scenario. In each room, specific cues of craving are displayed. These cues are not only visual, but also audio, emotional and socio-environmental. A central hall connects the other rooms and serves as a safe place for debriefing, where measures such as craving are assessed.
  Other Names: the use of the scenario in VR

SUMMARY:
Food craving is a major therapeutic issue in Eating Disorders with binge eating: the Bulimia Nervosa and the Binge Eating Disorder (BED). Food craving is linked to compulsive eating and its apprehension is currently based on classic Cognitive and Behavioural Therapies (CBT). However, it remains difficult to induce in therapy and a significant number of patients do not respond to classic CBTs. The development of exposure scenarios for CBT in virtual reality (VR) has allowed a gain in efficacy and in particular therapeutic effects lasting longer after treatment. Nevertheless, the stimuli used are often simple food visuals and insufficiently consider the many factors influencing food craving (physical, psychological, socio-environmental...) and VR immersion is still limited by the use of 3D laptops (fixed) rather than wireless headsets.

DETAILED DESCRIPTION:
Eating Disorders-specialized clinicians from Saint-Etienne University Hospital Center (CHU) and VR-specialized engineers from National School of Engineering of Saint-Etienne (ENISE) therefore collaborated in the creation of ReVBED, a VR-based exposure scenario for CBT for the induction of food craving in eating disorders with binge eating. ReVBED offers successive exposures to multimodal stimuli in a coherent scenario and in an immersive virtual environment via a wireless VR headset.

Our first objective is to validate the effectiveness of our scenario in inducing food craving in patients with bulimia and BED.

ELIGIBILITY:
Inclusion Criteria:

* Patients: who meet Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria for Bulimia Nervosa or Binge Eating Disorder
* Controls: paired to patients on age and level of education

Exclusion Criteria:

* Patients and controls:
* Under legal protection measure (guardianship, curatorship or safeguard of justice)
* Having a treatment being established and / or not stabilized (declarative) able to alter the physiological data recorded and the answers to the self-questionnaires
* Having one or more sensory deficit(s) or disorder(s) incompatible with the use of VR equipment (declarative)
* Patients: who have already benefited from specific care targeting food craving (declarative) Controls: with a score greater than or equal to 88 on the Bulimia Test (BULIT)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Verbal Rating Scales of food craving (VRS) | Change from the first exploration of virtual rooms to the last exploration (20 minutes)
  Evaluate variation in food craving assessed by Verbal Rating Scales (VRS) : self-assessment from 0 to 10 with 0 = "no food craving felt" and 10 = "maximum food craving felt")

SECONDARY OUTCOMES:
Verbal Rating Scales of food craving (VRS) | Change from the start of exploration of each virtual rooms to the end (5 minutes)
  Evaluate variation in food craving assessed by Verbal Rating Scales (VRS : self-assessment from 0 to 10 with 0 = "no food craving felt" and 10 = "maximum food craving felt")
Heart rate variation | Change from the first exploration of virtual rooms to the last exploration (20 minutes)
  Measurement of cyclical fluctuations with sensor
Pupillometry | Change from the first exploration of virtual rooms to the last exploration (20 min)
  Measurement of phase fluctuations of pupil diameters with visual sensor
Electro-Dermal Activity | Change from the first exploration of virtual rooms to the last exploration (20 minutes)
  Measurement of skin conductance fluctuations by amplifying the potential differences between two electrodes in contact with the subject's skin
Heart rate variation | Change from the start of exploration of each virtual rooms to the end (5 minutes)
  Measurement of cyclical fluctuations with sensor
Pupillometry | Change from the start of exploration of each virtual rooms to the end (5 minutes)
  Measurement of phase fluctuations of pupil diameters with visual sensor
Electro-Dermal Activity | Change from the start of exploration of each virtual rooms to the end (5 minutes)
  Measurement of skin conductance fluctuations by amplifying the potential differences between two electrodes in contact with the subject's skin
Variations of the measurements VRS of the food craving and each of the physiological measurements of the food craving | Change from the start of exploration of each virtual rooms to the end (5 minutes)
  Correlation between the variations of the VRS measurements and each of the physiological measurements (HRV, pupillometry and EDA) of the food craving induced in patients with bulimia and BED, compared to matched healthy controls.
Verbal Rating Scales of anxiety (VRS) | Change from the first exploration of virtual rooms to the last exploration (20 minutes)
  Evaluate variation of anxiety assessed by Verbal Rating Scales (VRS : self-assessment from 0 to 10 with 0 = "no food craving felt" and 10 = "maximum food craving felt")
Verbal Rating Scales of anxiety (VRS) | Change from the start of exploration of each virtual rooms to the end (5 minutes)
  Evaluate variation of anxiety assessed by Verbal Rating Scales (VRS) : self-assessment from 0 to 10 with 0 = "no food craving felt" and 10 = "maximum food craving felt")
Variations of the VRS food craving and of the VRS anxiety of the food craving | Change from the start of exploration of each virtual rooms to the end (5 minutes)
  Correlation between the variations Food Craving Verbal Rating Scales and Anxiety Verbal Rating Scales (VRS : self-assessment from 0 to 10 with 0 = "no felt" and 10 = "maximum felt") the VRS food craving and VRS anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Aurélia GAY, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No